CLINICAL TRIAL: NCT02825771
Title: Caring Contacts: A Strength-based, Suicide Prevention Trial in 4 Native Communities
Acronym: CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: University of Washington (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lonnie Nelson, Associate Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UWashington; 1R01MH106419-01A1 (NIH)
Record Dates: First submitted 2016-07-03; First posted 2016-07-07 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Suicidal Ideation; Suicide, Attempted
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care + Caring Contacts messages (Experimental): Usual care services plus caring contacts messages
  Interventions: Behavioral: Caring Contacts Messages; Behavioral: Usual Care
- Usual Care (Active Comparator): Usual care services provided in that community following identification of suicidal ideation or behavior.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Caring Contacts Messages — Text messages expressing care and support are sent following initial meeting on the following schedule: next day, 6 weekly, 9 bi-weekly, 7 monthly; one each on birthday, holiday, and seasonal (total of 25)
  Arms: Usual Care + Caring Contacts messages
Behavioral: Usual Care — Usual care consists of services available to the participant in their community to reduce their suicide risk and improve their behavioral health

SUMMARY:
Suicide is the second leading cause of death for American Indians and Alaska Natives aged 18 years and older. This study will evaluate Caring Contacts, a low-cost, sustainable intervention for suicide prevention that sends caring messages to people at risk. The investigators will implement the intervention at four tribal sites, leveraging community strengths and values to address this tragic health disparity in an underserved minority population.

DETAILED DESCRIPTION:
High rates of suicide are endemic in American Indian and Alaska Native (AI/AN) young adults. A recent study found that rates for young AI/AN adults in the Northern Plains and in Alaska are more than 4 times higher than for Whites of the same age in the same regions. Building social connections is a key goal of suicide prevention. One validated theoretical model asserts that belonging to a group is a fundamental human need. When this need is thwarted by social isolation or inadequate social support, a desire for death emerges. Studies of suicide prevention in AI/ANs underscore the cultural importance of connection to friends, family, caring neighbors, and community leaders. These traditions of community cohesion can be leveraged to protect young AI/AN adults against suicidal ideation and behavior. Caring Contacts is a suicide prevention program that supplements standard care by promoting human connectedness. People at risk for suicide often lose contact with the healthcare system and receive no follow-up care. For one year after initial contact, Caring Contacts seeks out such individuals to send messages expressing care, concern, and interest. It is the only intervention shown to prevent suicide in any population in a randomized, controlled trial. Based on a two year collaborative process with four tribal partners as part of a pilot grant, this study will evaluate a locally feasible, culturally appropriate Caring Contacts intervention that will use text messaging, email, and postal mail. This study uses a randomized, controlled trial (RCT) to evaluate this approach to suicide prevention in 1,200 high-risk AI/ANs aged 18 and older from our four partner communities. Specific Aims are to: 1) Compare the effectiveness of usual care (control) to the control condition plus caring text messages (intervention) for reducing suicidal ideation, suicide attempts, and suicide related hospitalizations. 2) Evaluate social connectedness as a mediating factor for the effect of Caring Contacts via text message on suicidality. The US Surgeon General's National Strategy for Suicide Prevention identifies connectedness to others as a primary protective factor against suicidality. By adapting and disseminating the Caring Contacts approach, which has demonstrated effectiveness in non-Native populations, this study will evaluate a low-cost, sustainable intervention for addressing the profound disparity of suicide risk experienced by young adult AI/ANs.

ELIGIBILITY:
Inclusion Criteria:

1. be suicidal (Suicidal Ideation Questionnaire clinical cut-off score ≥ 32) or have a documented or self-reported suicide attempt within the past year
2. be 18 years or older
3. self-identify as American Indian or Alaska Native
4. are willing to be contacted periodically via text, email, or postal mail
5. able to participate voluntarily
6. speak and read English

Exclusion Criteria:

1) Cognitively unable and willing to independently provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation Questionnaire (SIQ) | 12 and 18 months
  The SIQ comprises 15 items assessing frequency of suicidal thoughts in the past month
Suicide Attempt and Self-Injury Count (SASI-Count) | 12 and 18 months
  The SASI-Count interview assesses the method, intent, treatment received, and lethality for all suicide attempts in the follow-up time frame
Suicide-related hospitalizations | 12 and 18 months
  Hospitalizations will be assessed using the American Indian Services Utilization and Psychiatric Epidemiology Risk and Protective Factors Project (AI-SUPERPFP) measure of service utilization which captures all admissions to inpatient medical and psychiatric care as well as emergency room visits

SECONDARY OUTCOMES:
Interpersonal Needs Questionnaire (INQ) Thwarted Belongingness subscale | 12 and 18 months
  Thwarted belongingness is one of two subscales on the INQ that measures the lack of perceived social connectedness

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie A Nelson, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Collaborative decision with four tribal partners.

REFERENCES:
- [Derived] Hebert LE, Fruhbauerova M, Evanson A, Bogic M, Petras A, Shaw J, Muller CJ, Nelson L, Comtois KA. Caring Texts, a strength-based, suicide prevention trial in 5 native communities: Research design and methods. Contemp Clin Trials. 2022 Dec;123:106966. doi: 10.1016/j.cct.2022.106966. Epub 2022 Oct 14. PMID 36252937